CLINICAL TRIAL: NCT03280628
Title: A Randomized Controlled Trial Comparing Cosmetic Outcomes of Pediatric Laceration Closure Using a Tissue Adhesive (Dermabond™) Versus Adhesive Strips (Steri-Strips™) Versus Absorbable Sutures
Brief Title: Trial Comparing Cosmetic Outcomes of Pediatric Laceration Closure Using Skin Glue, Medical Tape Versus Stitches
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID-19 pandemic made prospective enrollment no longer possible
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Holly Hanson, Asst Professor of Clinical Pediatrics, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 171108
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2022-09

CONDITIONS: Laceration
MeSH Terms: conditions — Lacerations | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Plastic Surgeons who rate all scars at the end of the study are blinded to the closure method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Absorbable Sutures (Active Comparator): Patients will have their laceration closed with sutures that absorb on their own and do not need to be removed.
  Interventions: Procedure: Absorbable Sutures
- Steri-Strips (Experimental): Patients will have their laceration closed with a special medical tape called "Steri-Strips."
  Interventions: Procedure: Steri-Strips
- Dermabond (Experimental): Patients will have their laceration closed with a special skin glue called "Dermabond"
  Interventions: Procedure: Dermabond

INTERVENTIONS:
Procedure: Absorbable Sutures — The patient's doctor will close the patient's laceration with absorbable sutures.
  Other Names: Stitches
  Arms: Absorbable Sutures
Procedure: Steri-Strips — The patient's doctor will close the patient's laceration with Steri-Strips.
  Other Names: Medical tape
  Arms: Steri-Strips
Procedure: Dermabond — The patient's doctor will close the patient's laceration with Dermabond.
  Other Names: Skin glue
  Arms: Dermabond

SUMMARY:
There are several methods of closing a skin cut: stitches, skin glue, and medical tape. Stitches have been used for a long time to close skin cuts. Skin glue (invented in the 1970s) and medical tape (invented in the 1960s) are two newer methods to close skin cuts. The purpose of this study is to find out which method (stitches, skin glue, or medical tape) of closing skin cuts results in the least amount of scarring. Other things the investigators will be looking at are which method is the cheapest, which causes the least pain, which requires the least amount of sedation, and which method patients and parents like the best.

DETAILED DESCRIPTION:
When a child comes in to the Emergency Room with a skin cut, if the child and their parents consent to being in the study, they will be randomly assigned to one of three groups: stitches, skin glue, or medical tape. There will be about 30 kids in each group, and thus a goal of 90 kids total in the study.

In the Emergency Room, a lidocaine ointment will be placed on the child's cut to decrease pain. The cut will be cleaned out with sterile saline. Then, depending on which method is used, the cut will be closed with either stitches, skin glue, or medical tape by their doctor. The participants will be asked to answer a short questionnaire. Finally, they will be given discharge instructions and sent home. At 3 months, the investigators will call parents for a quick questionnaire over the phone and parents will be asked to take a picture of the patient's scar and send it to the study staff.

Once all 90 pictures have been collected, two Plastic Surgeons will be asked to rate the scars in terms of how they look. The Plastic Surgeons will not know which method was used to close which cut. Once all of the scars have been rated, the averages of scars will be compared for each closure method. The investigators will also look at how much each method cost, how much extra pain medications or sedation each group used, and which method was liked best.

ELIGIBILITY:
Inclusion Criteria:

* Medical complaint of laceration
* Single, linear laceration
* Laceration less than 5 cm in length and 0.5 cm in width
* Laceration less than 12 hours old
* Laceration minimally contaminated (no visible dirt in wound)
* Parents and child speak English

Exclusion Criteria:

* Significant medical history that may impact wound healing (hematologic or oncologic diagnosis requiring chemotherapy, ichthyosis, epidermolysis bullosa, etc.)
* Use of oral steroids (more than 5 days in the past month)
* History of keloid formation
* Allergy to skin glue, medical tape, or topical anesthetics
* Lacerations requiring deep sutures
* Lacerations caused by animal bites or scratches
* Lacerations located on the scalp, eyebrow, eyelid, lip, mucosa, joint or nail bed
* No access to photographic capabilities (camera or smartphone) and/or e-mail, OR unable to return to the Vanderbilt Children's Hospital Emergency Room to have a picture taken at 3 months

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2017-09-23 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly R Hanson, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barton MS, Chaumet MSG, Hayes J, Hennessy C, Lindsell C, Wormer BA, Kassis SA, Ciener D, Hanson H. A Randomized Controlled Comparison of Guardian-Perceived Cosmetic Outcome of Simple Lacerations Repaired With Either Dermabond, Steri-Strips, or Absorbable Sutures. Pediatr Emerg Care. 2024 Oct 1;40(10):700-704. doi: 10.1097/PEC.0000000000003244. Epub 2024 Aug 2. PMID 39141836

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Started | 20 | 17 | 18
Completed | 12 | 11 | 7
Not Completed | 8 | 6 | 11
Not completed — Lost to Follow-up | 8 | 6 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond | Total
Number analyzed (Participants) | 20 | 17 | 18 | 55
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.50 [2.75 to 5.00] | 3.00 [2.00 to 5.00] | 4.00 [3.00 to 5.00] | 3.00 [2.75 to 5.00]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 12
  Male | 17 | 12 | 14 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 18 | 16 | 16 | 50
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 4 | 12
  White | 14 | 12 | 10 | 36
  More than one race | 1 | 1 | 3 | 5
  Unknown or Not Reported | 0 | 1 | 1 | 2
Laceration Length (cm) [Median (Inter-Quartile Range); unit: cm] | 1.50 [1.19 to 2.00] | 1.00 [1.00 to 1.50] | 1.50 [1.00 to 2.00] | 1.50 [1.00 to 1.94]
Laceration Width (cm) [Median (Inter-Quartile Range); unit: cm] | 0.50 [0.30 to 0.50] | 0.50 [0.30 to 0.50] | 0.50 [0.50 to 0.50] | 0.50 [0.30 to 0.50]
Training Level of Proceduralist [Count of Participants; unit: Participants]
  Resident | 7 | 11 | 10 | 28
  Fellow | 4 | 2 | 1 | 7
  Nurse Practitioner | 6 | 3 | 4 | 13
  Attending | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Cosmetic Outcome of Scar at 3 Months
Description: Two blinded Plastic Surgeons will rate the cosmetic outcome of the laceration using a 0 to 100 mm Visual Analogue Scale with a score of 0 corresponding to "worst scar" and a score of 100 corresponding to "best scar"
Time Frame: 3 months
Population: 55 subjects were enrolled in the Emergency Department but only 30 subjects sent 3 month follow-up photos of their child's scar thus only 30 scars were reviewed by the plastic surgeons.
Measure: Median (Inter-Quartile Range); unit: units on a visual analog scale
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Number analyzed (Participants) | 12 | 11 | 7
units on a visual analog scale | 64.00 [51.00 to 76.00] | 54.00 [35.50 to 66.75] | 48.50 [29.50 to 78.75]

2. Secondary Outcome: Pain Experienced by Patient as Reported by Parent
Description: Parents will each be asked to score how much pain they felt the patient experienced using a 100 mm Visual Analogue Scale with a score of 0 corresponding to "No pain" and a score of 100 corresponding to "Terrible pain."
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Number analyzed (Participants) | 20 | 17 | 18
units on a scale | 17.00 [1.50 to 51.50] | 22.00 [9.00 to 28.00] | 11.00 [3.00 to 24.50]

3. Secondary Outcome: Satisfaction With Time in the Emergency Department
Description: Parents will report their satisfaction with Emergency Department length of stay using a 100-point visual analog scale with "100" meaning completely satisfied and "0" meaning not at all satisfied
Time Frame: Baseline to wound closure, up to 30 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Number analyzed (Participants) | 20 | 17 | 18
units on a scale | 89.50 [45.25 to 98.50] | 92.00 [83.00 to 100.00] | 94.00 [71.25 to 100.00]

4. Secondary Outcome: Likelihood That Parent Would Recommend Laceration Closure Method
Description: Parents will be asked to rate how likely they would be to recommend the closure method used for their child using a 0 to 100 mm Visual Analogue Scale with a score of 0 corresponding to "Extremely unlikely" and a score of 100 corresponding to "Extremely likely"
Time Frame: Post-wound closure, approximately 30 minutes
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Number analyzed (Participants) | 20 | 17 | 18
units on a scale | 99.50 [88.00 to 100.00] | 99.00 [95.00 to 100.00] | 99.50 [94.50 to 100.00]

5. Secondary Outcome: Number of Complications of the Wound Site
Description: Parents will be asked by phone at 3 months if there were any complications with their child's cut (infection, opening of the wound, etc.). Investigators will count the number of complications reported.
Time Frame: 3 months
Population: 55 subject were enrolled but only 30 completed 3 month follow-up. This outcome measure was collected at 3 months.
Measure: Number; unit: complications
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Number analyzed (Participants) | 12 | 11 | 7
complications | 0 | 0 | 0

6. Secondary Outcome: Parental Reported Satisfaction With the Cosmetic Appearance of the Scar
Description: Parents will rate the cosmetic outcome of the laceration using a 0 to 100 mm Visual Analogue Scale with a score of 0 corresponding to "worst scar" and a score of 100 corresponding to "best scar".
Time Frame: 3 months
Population: Only 30 parents/subjects provided 3 month follow-up photos of their scar
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Number analyzed (Participants) | 12 | 11 | 7
units on a scale | 70.50 [59.75 to 76.75] | 67.00 [55.00 to 78.00] | 85.00 [73.00 to 90.00]

7. Secondary Outcome: Presence of Train Tracks at the Scar Site
Description: Plastic Surgeons will record if a scar appears to have "train tracks" (or small dots on either side of a scar, all along the scar, usually caused by stitches) as they are rating each photo of the scar at 3 months post-closure. Surgeons will answer "yes" or "no".
Time Frame: 3 months
Population: 55 subjects were enrolled but only 30 subjects submitted scar photos 3 months after closure.
Measure: Number; unit: scars with train tracks
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
Number analyzed (Participants) | 12 | 11 | 7
scars with train tracks | 4 | 4 | 3

ADVERSE EVENTS:
Time Frame: Baseline to 3 months post-procedure.
Description: No difference in definition for adverse event and serious adverse event.
Arm/Group | Absorbable Sutures | Steri-Strips | Dermabond
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/18

LIMITATIONS AND CAVEATS:
Early termination of the study due to limitation regarding the COVID-19 pandemic and prospective enrollment of pediatric patients in the Emergency Department. There were also only 55% of subjects who performed 3 month follow-up thus our primary outcome can only be measured on these subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT03280628/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT03280628/ICF_001.pdf